CLINICAL TRIAL: NCT06316154
Title: Presentation of Protoscolexes and Acephalocysts in the Fibrous Capsule Area of the Liver With Echinococcosis During Organ-preserving Surgery
Brief Title: Presentation of Protoscolexes and Acephalocysts in the Fibrous Capsule Area of the Liver With Echinococcosis
Acronym: PAFCLE
Status: Recruiting | Type: Observational
Sponsor: Republican Specialized Scientific and Practical Medical Center of Surgery Named After V. Vakhidov (Other)
Responsible Party: Principal Investigator, Azam Babadjanov, Professor, Republican Specialized Scientific and Practical Medical Center of Surgery Named After V. Vakhidov
Other Study IDs: 12032024
Record Dates: First submitted 2024-03-12; First posted 2024-03-18 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-09

CONDITIONS: Echinococcosis, Hepatic
MeSH Terms: conditions — Echinococcosis, Hepatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Echinococcectomy — Echinococcectomy with subsequent pathomorphological analysis of liver parenchyma next to and in the thickness of the fibrous capsule

SUMMARY:
The objective of the study is to determine the presence of germinal elements of echinococcosis in the liver parenchyma next to and in the thickness of the fibrous capsule of hydatid cysts.

ELIGIBILITY:
Inclusion Criteria:

* Presence of primary or recurrent liver echinococcosis disease requiring surgical treatment
* Cyst diametr >5 cm;
* Performing one of the surgical treatment of liver echinococcosis with intraoperative sampling of part of the fibrous capsule with or without adjacent liver tissue for research;
* Signed informed consent of patients for inclusion in the study;

Exclusion Criteria:

* Liver echinococcosis with cysts less than 5 cm in diametr;
* Presence of severe concomitant disorders

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary or recurrent liver echinococcosis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-10-22 (Actual); Primary Completion 2026-12-22 (Estimated); Study Completion 2026-12-25 (Estimated)

PRIMARY OUTCOMES:
Presence of viable germinal elements of echinococcosis | 1 day
  Identification of viable germinal elements of echinococcosis according to morphological analysis

SECONDARY OUTCOMES:
Recurrence of liver echinococcosis | 1 year
  Identification of frequency of liver echinococcosis in postoperative period

CONTACTS AND LOCATIONS:
Locations (1):
- Republican specialized scientific and practical medical center of surgery named after academician V.Vakhidov, Tashkent, Uzbekistan, Uzbekistan

IPD SHARING:
Plan to Share IPD: No